CLINICAL TRIAL: NCT01466179
Title: An Open Label, Multicenter, Phase II Study to Evaluate Efficacy and Safety of the BiTE® Antibody Blinatumomab in Adult Patients With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia (ALL)
Brief Title: Clinical Study With Blinatumomab in Patients With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen Research (Munich) GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT103-211; 2011-002257-61 (EudraCT Number)
Record Dates: First submitted 2011-10-28; First posted 2011-11-07 (Estimated); Results first posted 2015-01-22 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: B-ALL; relapsed ALL; refractory ALL; adult ALL; Leukemia; Leukemia, Lymphoid; precursor cell lymphoblastic leukemia-lymphoma; Lymphatic diseases; Lymphoproliferative disorders; bispecific antibody; anti-CD19; Immunotherapeutic treatment; immunoproliferative disorders
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Leukemia, Lymphoid; Lymphatic Diseases; Lymphoproliferative Disorders; Immunoproliferative Disorders | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blinatumomab (Experimental): Participants received blinatumomab by continuous intravenous (CIV) infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The initial dose was 9 μg/day for the first seven days of treatment, escalated to 28 μg/day starting from Week 2 of treatment.
  Interventions: Biological: Blinatumomab

INTERVENTIONS:
Biological: Blinatumomab — Continuous intravenous infusion over four weeks per treatment cycle
  Other Names: AMG103; MT103; BLINCYTO™

SUMMARY:
The purpose of this study is to confirm whether the bispecific T cell engager antibody blinatumomab (MT103) is effective and safe in the treatment of patients with relapsed or refractory Acute Lymphoblastic Leukemia (ALL).

DETAILED DESCRIPTION:
Relapsed/refractory B-precursor ALL in adult patients is an aggressive malignant disease with dismal prognosis. Several studies have reported long term survival to be below 10%. Major prognostic factors are duration of first complete remission (CR1) and age. With current salvage chemotherapy, complete remission (CR) rate is low (20 to 30%) in patients in first salvage with short duration (< one year) of first remission, patients relapsed after first salvage, or patients aged 60 years and older. Duration of CR is usually very short (median disease free survival [DFS]: 2.0-7.5 months). Allogeneic hematopoietic stem cell transplantation (HSCT) may provide a curative treatment option for patients in CR with a satisfactory donor and appropriate clinical status including age, organ function, and remission status. Allogeneic HSCT is not an option in most elderly patients with relapsed ALL. Additional therapeutic approaches are urgently needed.

Blinatumomab is a bispecific single-chain antibody derivative against CD (cluster of differentiation)19 and CD3, designed to link B cells and T cells resulting in T cell activation and a cytotoxic T cell response against CD19-expressing cells. In vitro data indicate CD19+ lymphoma and leukemia cell lines to be extremely sensitive to blinatumomab-mediated cytotoxicity. Blinatumomab has the potential to provide meaningful therapeutic benefits to patients compared with existing treatments for this patient population.

This study consists of a screening period, a treatment period and a follow-up period. Participants receive one to five treatment cycles of blinatumomab at a target dose of 28 μg/day. In the first cycle, the initial dose is 9 μg/day for the first seven days of treatment, escalated to 28 μg/day starting from Week 2 of treatment.

Participants who achieve remission within two cycles of treatment can receive up to three additional cycles of consolidation treatment or proceed to allogeneic HSCT. In the event of progression or relapse within the treatment period, treatment will be terminated. Participants with hematological relapse during the efficacy or safety follow-up period may receive up to three additional cycles of blinatumomab (retreatment) for a maximal total of eight cycles at the investigator´s discretion.

Thirty days after end of the last treatment, participants have an end-of-core-study visit. Following this, there are efficacy follow-up visits at 3, 6, 9, 12, 18 and 24 months at the most after treatment start. Once efficacy follow-up is complete, information on survival collected at least every six months until death or at least until three years after treatment start, whichever occurs earlier (survival follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Philadelphia chromosome (Ph)-negative B-precursor ALL, with any of the following:

  * relapsed or refractory with first remission duration less than or equal to 12 months in first salvage or
  * relapsed or refractory after first salvage therapy or
  * relapsed or refractory within 12 months of allogeneic hematopoietic stem cell transplantation (HSCT)
* 10% or more blasts in bone marrow
* In case of clinical signs of additional extramedullary disease: measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Age ≥ 18 years

Exclusion Criteria:

* Patients with Ph-positive ALL
* Patients with Burkitt's Leukemia according to World Health organization (WHO) classification
* History or presence of clinically relevant central nervous system (CNS) pathology
* Active ALL in the CNS or testes
* Current autoimmune disease or history of autoimmune disease with potential CNS involvement
* Autologous HSCT within six weeks prior to start of blinatumomab treatment
* Allogeneic HSCT within three months prior to start of blinatumomab treatment
* Any active acute graft versus-host disease (GvHD), or active chronic GvHD Grade 2 - 4
* Any systemic therapy against GvHD within two weeks prior to start of blinatumomab treatment
* Cancer chemotherapy within two weeks prior to start of blinatumomab treatment
* Radiotherapy within two weeks prior to start of blinatumomab treatment
* Immunotherapy (e.g., rituximab) within four weeks prior to start of blinatumomab treat-ment
* Any investigational anti-leukemic product within four weeks prior to start of blinatumomab treatment
* Treatment with any other investigational medicinal product (IMP) after signature of informed consent
* Eligibility for allogeneic HSCT at the time of enrollment
* Known hypersensitivity to immunoglobulins or to any other component of the IMP formulation
* Abnormal laboratory values indicative of inadequate renal or liver function
* History of malignancy requiring treatment other than ALL within five years prior to start of blinatumomab treatment with the exception of basal cell or squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix
* Any concurrent disease or medical condition that is deemed to interfere with the conduct of the study
* Infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus or hepatitis C virus
* Pregnant or nursing women
* Women of childbearing potential not willing to use an effective form of contraception. Male patients not willing to ensure not to beget a child
* Previous treatment with blinatumomab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Gökbuget, MD, Principal Investigator — Klinikum der Goethe Universität Frankfurt; Max Topp, MD, Principal Investigator — Julius-Maximilians-Universität, Medizinische Klinik und Poliklinik II, Würzburg; Hagop Kantarjian, MD, Principal Investigator — MD Anderson Cancer Center, Houston, Texas
Locations (39):
- United States (12):
  - City of Hope, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Dana Farber Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Streets, Buffalo, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- France (4):
  - CHU d'Angers, Angers
  - Hôpital de l'hôtel Dieu, Nantes
  - Hôpital Saint Louis, Paris
  - CHU de Purpan, Toulouse
- Germany (9):
  - Charité - Campus Benjamin Franklin, Berlin
  - Klinikum der Goethe Universität, Medizinische Klinik II, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Julius-Maximilians-Universität, Medizinische Klinik und Poliklinik II, Würzburg
- Italy (6):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Azienda Ospedaliera Antonio Cardarelli, Naples
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - Università La Sapienza di Roma, Rome
  - Azienda Ospedaliero-Universitaria, Turin
  - Azienda Ospedaliera di Verona, Verona
- Spain (5):
  - ICO Hospital Germans Trias I Pujol, Badalona
  - Hospital Clínic Servei d´Hematologia, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
- United Kingdom (3):
  - University Hospitals Bristol NHS, Bristol
  - Royal Free Hampstead NHS Trust, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- [Derived] Gokbuget N, Kantarjian HM, Bruggemann M, Stein AS, Bargou RC, Dombret H, Fielding AK, Heffner L, Rigal-Huguet F, Litzow M, O'Brien S, Zugmaier G, Gao S, Nagorsen D, Forman SJ, Topp MS. Molecular response with blinatumomab in relapsed/refractory B-cell precursor acute lymphoblastic leukemia. Blood Adv. 2019 Oct 22;3(20):3033-3037. doi: 10.1182/bloodadvances.2019000457. PMID 31648325
- [Derived] Zhu M, Kratzer A, Johnson J, Holland C, Brandl C, Singh I, Wolf A, Doshi S. Blinatumomab Pharmacodynamics and Exposure-Response Relationships in Relapsed/Refractory Acute Lymphoblastic Leukemia. J Clin Pharmacol. 2018 Feb;58(2):168-179. doi: 10.1002/jcph.1006. Epub 2017 Sep 18. PMID 28922466
- [Derived] Barlev A, Lin VW, Katz A, Hu K, Cong Z, Barber B. Estimating Long-Term Survival of Adults with Philadelphia Chromosome-Negative Relapsed/Refractory B-Precursor Acute Lymphoblastic Leukemia Treated with Blinatumomab Using Historical Data. Adv Ther. 2017 Jan;34(1):148-155. doi: 10.1007/s12325-016-0447-x. Epub 2016 Nov 21. PMID 27873237
- [Derived] Zhu M, Wu B, Brandl C, Johnson J, Wolf A, Chow A, Doshi S. Blinatumomab, a Bispecific T-cell Engager (BiTE((R))) for CD-19 Targeted Cancer Immunotherapy: Clinical Pharmacology and Its Implications. Clin Pharmacokinet. 2016 Oct;55(10):1271-1288. doi: 10.1007/s40262-016-0405-4. PMID 27209293
- [Derived] Topp MS, Gokbuget N, Stein AS, Zugmaier G, O'Brien S, Bargou RC, Dombret H, Fielding AK, Heffner L, Larson RA, Neumann S, Foa R, Litzow M, Ribera JM, Rambaldi A, Schiller G, Bruggemann M, Horst HA, Holland C, Jia C, Maniar T, Huber B, Nagorsen D, Forman SJ, Kantarjian HM. Safety and activity of blinatumomab for adult patients with relapsed or refractory B-precursor acute lymphoblastic leukaemia: a multicentre, single-arm, phase 2 study. Lancet Oncol. 2015 Jan;16(1):57-66. doi: 10.1016/S1470-2045(14)71170-2. Epub 2014 Dec 16. PMID 25524800

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to adult patients with relapsed / refractory B-precursor acute lymphoblastic leukemia (ALL).
  The study protocol originally used a Simon 2-stage design and was subsequently expanded to include a third stage. Protocol amendment 4 added an additional cohort of participants for central nervous system evaluations.
Pre-assignment Details: Two hundred twenty-five participants enrolled in the study overall. Results below include data for 189 participants enrolled in the first 3 stages of the study (the primary analysis set). An additional 36 participants enrolled in the Additional Evaluation Cohort are not reported here as the study is ongoing and data collection has not completed.
Period: Overall Study
Arm/Group | Blinatumomab
Started | 189 (Participants enrolled during the first 3 stages of the study)
Completed | 10 (Completed 5 cycles of treatment; Data as of the time of the data cut-off date (10 October 2013).)
Not Completed | 179
Not completed — Ongoing in core study | 2
Not completed — Physician Decision | 46
Not completed — Progressive disease | 43
Not completed — Adverse Event | 32
Not completed — Disease relapse | 23
Not completed — Lack of Efficacy | 14
Not completed — Death | 7
Not completed — Withdrawal by Subject | 7
Not completed — Protocol Violation | 2
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: Primary Analysis Set
Arm/Group | Blinatumomab
Number analyzed (Participants) | 189
Age, Continuous [Median (Full Range); unit: years] | 39.0 [18 to 79]
Age, Customized [Number; unit: participants]
  18 to < 35 years | 90
  35 to < 55 years | 46
  55 to < 65 years | 28
  ≥ 65 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 119
Race/Ethnicity, Customized [Number; unit: participants] — Race was not permitted to be collected in France
  participants
    White | 145
    Asian | 6
    Black or African American | 7
    American Indian or Alaska native | 1
    Native Hawaiian or other Pacific Islander | 1
    Other | 9
    Not recorded | 20
Disease stage entry criteria met [Number; unit: participants] — HSCT = hematopoietic stem cell transplantation
  participants
    Primary refractory | 16
    Relapse ≤ 12 months of allogeneic HSCT | 39
    Entering first salvage; first remission ≤ 12 mo | 23
    Entering second or greater salvage therapies | 108
    No criteria met | 3
Number of prior relapses [Number; unit: participants]
  0 | 16
  1 | 107
  2 | 46
  >2 | 20
Prior allogeneic HSCT and prior relapses [Number; unit: participants] — alloHSCT = allogeneic hematopoietic stem cell transplantation
  participants
    Prior allogeneic HSCT | 64
    No prior alloHSCT, no prior relapse | 16
    No prior alloHSCT, 1 prior relapse | 84
    No prior alloHSCT, 2 prior relapses | 22
    No prior alloHSCT, > 2 prior relapses | 3
Number of prior salvage therapies [Number; unit: participants]
  No prior salvage therapy | 38
  1 prior salvage therapy | 77
  2 prior salvage therapies | 42
  > 2 prior salvage therapies | 32
Time since initial diagnosis [Median (Full Range); unit: months] | 16.59 [1.9 to 249.0]
Time since last relapse [Median (Full Range); unit: months] — Reported for 173 participants with a prior relapse (the other16 participants were primary refractory with no prior relapses).
  months | 1.38 [0.1 to 56.8]
Baseline bone marrow blast category [Number; unit: participants] — Bone marrow blasts were assessed by local and central laboratories; reported data are based on maximum central and local laboratory assessments.
  participants
    < 10% | 1
    10% - < 50% | 43
    ≥ 50% | 145

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Best Response of Complete Remission or Complete Remission With Only Partial Hematological Recovery Within 2 Cycles of Treatment
Description: Hematological assessments were performed from bone marrow biopsy samples. All hematological assessments of bone marrow were reviewed in a central reference laboratory.
  Hematological remissions were defined by the following criteria:
  Complete Remission (CR):
  * bone marrow blasts ≤ 5%
  * no evidence of disease
  * full recovery of peripheral blood counts:
    * platelets > 100,000/μL, and
    * absolute neutrophil count (ANC) > 1,000/μL
  Complete Remission With Partial Hematological Recovery (CRh*):
  * bone marrow blasts ≤ 5%
  * no evidence of disease
  * partial recovery of peripheral blood counts:
    * platelets > 50,000/μL, and
    * ANC > 500/μL.
Time Frame: Within the first 2 cycles of treatment, 12 weeks
Population: The Primary Analysis Set (PAS), defined as participants from the first 3 stages of the study who received any infusion of blinatumomab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 189
percentage of participants | 42.9 [35.7 to 50.2]

2. Secondary Outcome: Time to Hematological Relapse (Duration of Response)
Description: Time to hematological relapse was measured for participants in remission during the core study (the time from the first infusion through 30 days after the last infusion), from the time the participant first achieved remission until first documented relapse or death due to disease progression. Participants without documented relapse (hematological or extramedullary) and who did not die were censored at the time of their last bone marrow assessment or their last survival follow-up visit confirming remission. Participants who died without having reported hematological relapse or without showing any clinical sign of disease progression were censored on their date of death.
  Hematological relapse is defined as:
  * proportion of blasts in bone marrow > 5% after documented CR/CRh* or
  * blasts in peripheral blood after documented CR/CRh*.
  Time to hematological relapse was analyzed by Kaplan-Meier methods and the median observation time was calculated by the reverse Kaplan Meier method.
Time Frame: Up to the data cut-off date of 10 October 2013; median observation time was 8.0 months.
Population: Participants who reached complete remission or complete remission with partial hematological recovery during the core study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 82
months | 6.7 [5.1 to NA] — Not estimable due to the number of events during the observation period.

3. Secondary Outcome: Percentage of Participants Who Received an Allogeneic Hematopoietic Stem Cell Transplant (HSCT) During Blinatumomab Induced Remission
Description: Participants who were eligible for allogeneic HSCT were those who achieved remission (complete response or complete response with partial recovery of peripheral blood counts) after 2 cycles of blinatumomab treatment, and no further anti-leukemic medication was given before HSCT.
Time Frame: Up to the data cut-off date of 10 October 2013. Maximum duration on study was 17.8 months.
Population: Participants who reached complete remission or complete remission with partial hematological recovery during the first 2 cycles of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 81
percentage of participants | 39.5 [28.8 to 51.0]

4. Secondary Outcome: Percentage of Participants With a Best Response of Complete Remission Within 2 Cycles of Treatment
Description: Complete Remission was defined by the following criteria:
  * bone marrow blasts ≤ 5%
  * no evidence of disease
  * full recovery of peripheral blood counts:
    * platelets > 100,000/μL, and
    * absolute neutrophil count (ANC) > 1,000/μL
Time Frame: Within the first 2 cycles of treatment, 12 weeks
Population: Primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 189
percentage of participants | 33.3 [26.7 to 40.5]

5. Secondary Outcome: Percentage of Participants With a Best Response of Complete Remission With Only Partial Hematological Recovery Within 2 Cycles of Treatment
Description: Complete Remission With Partial Hematological Recovery was defined by the following criteria:
  * bone marrow blasts ≤ 5%
  * no evidence of disease
  * partial recovery of peripheral blood counts:
    * platelets > 50,000/μL, and
    * ANC > 500/μL.
Time Frame: Within the first 2 cycles of treatment, 12 weeks
Population: Primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 189
percentage of participants | 9.5 [5.7 to 14.6]

6. Secondary Outcome: Percentage of Participants With a Best Response of Partial Remission Within 2 Cycles of Treatment
Description: Partial Remission is defined as bone marrow blasts 6% to 25% with at least a 50% reduction from baseline.
Time Frame: Within the first 2 cycles of treatment, 12 weeks
Population: Primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 189
percentage of participants | 2.6 [0.9 to 6.1]

7. Secondary Outcome: Relapse-free Survival
Description: Relapse-free survival was assessed for participants who achieved a complete remission or complete remission with partial hematological recovery during the core study and was measured from the time the participant first achieved remission until first documented relapse or death due to any cause. Participants without a documented relapse (hematological or extramedullary) or who did not die were censored at the time of their last bone marrow assessment or their last survival follow-up visit confirming remission.
  Relapse free survival was estimated using Kaplan-Meier methods and the median observation time was calculated by the reverse Kaplan Meier method.
Time Frame: Up to the data cut-off date of 10 October 2013; median observation time was 8.9 months.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 82
months | 5.9 [4.8 to 8.3]

8. Secondary Outcome: Event-free Survival
Description: Event-free survival was calculated from the start date of blinatumomab infusion until the date of bone marrow aspiration at which hematological relapse was first detected, or the date of diagnosis on which the hematological or extramedullary relapse was documented or the date of start of any new therapy for ALL (excluding HSCT), or the date of death, whichever was earlier. Participants who did not achieve complete remission or complete remission with partial hematological recovery during the core study were evaluated as having an event on Day 1. Participants in remission who did not experience hematological relapse, did not receive a new therapy for ALL (excluding HSCT), and did not die were censored on the date of the last available bone marrow aspiration or on the last date of survival follow-up visit, whichever was later.
  Event free survival was estimated using Kaplan-Meier methods and the median observation time was calculated by the reverse Kaplan Meier method.
Time Frame: Up to the data cut-off date of 10 October 2013; median observation time was 9.8 months.
Population: Primary analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 189
months | 0.0 [0.0 to 1.0]

9. Secondary Outcome: Overall Survival
Description: Overall survival was measured for all participants from the time the participant received the first treatment of blinatumomab until death due to any cause or the date of the last follow-up. Participants who did not die were censored on the last documented visit date or the date of the last phone contact when the patient was last known to have been alive. Overall survival was estimated using Kaplan-Meier methods. The median follow-up time with respect to overall survival was calculated by the reverse Kaplan Meier method.
Time Frame: Up to the data cut-off date of 10 October 2013; median observation time was 9.8 months.
Population: Primary analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Blinatumomab
Number analyzed (Participants) | 189
months | 6.1 [4.2 to 7.5]

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Adverse events (AEs) were evaluated for severity according to the the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4, as follows: Grade 1 - Mild AE; Grade 2 - Moderate AE; Grade 3 - Severe AE; Grade 4 - Life-threatening or disabling AE; Grade 5 - Death.
  The investigator used medical judgment to determine if there was a causal relationship (ie, related, unrelated) between an adverse event and blinatumomab.
  An AE was considered "serious" if it resulted in death, was life-threatening, requires or prolongs inpatient hospitalization, results in persistent or significant incapacity or substantial disruption to conduct normal life functions, is a congenital anomaly or birth defect or is a medically important condition.
  Progressive disease was not an adverse event, per the protocol, unless it was more severe than expected for the patient. Therefore, many deaths due to progressive disease were not counted as adverse events.
Time Frame: From the start of the first infusion to 30 days after the end of the last infusion in the core study or from the start of the first retreatment cycle infusion to 30 days after the end of the last retreatment cycle, median treatment duration was 42.2 days.
Population: Full analysis set (FAS), defined as all patients who received any infusion of blinatumomab.
Measure: Number; unit: participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 189
participants
  Any adverse event (AE) | 188
  Adverse events of at least CTC grade 3 | 155
  Treatment-related adverse events | 166
  Related adverse events of at least CTC grade 3 | 105
  Serious adverse events | 121
  Serious adverse events of at least CTC grade 3 | 105
  Related serious adverse events | 69
  AEs leading to interruption of blinatumomab | 63
  AEs leading to discontinuation of blinatumomab | 34
  Related AE leading to treatment discontinuation | 18
  AEs leading to death | 28
  Related AEs leading to death | 3

11. Secondary Outcome: 100-Day Mortality After Allogeneic Hematopoietic Stem Cell Transplant
Description: The analysis of 100-day mortality after allogeneic HSCT was assessed for all participants who received an allogeneic HSCT while in remission (CR/CRh*) following treatment with blinatumomab. 100-day mortality after allogeneic HSCT was calculated relative to the date of allogeneic HSCT.
  Patients alive were censored on the last documented visit date or the date of the last phone contact when the patient was last known to have been alive.
  The 100-day mortality rate after allogeneic HSCT was defined as the percentage of patients having died up to 100 days after allogeneic HSCT estimated using the estimated time to death in percent calculated by Kaplan-Meier methods.
Time Frame: From the date of allogeneic HSCT until the data cut-off date of 10 October 2013; median observation time was 7.4 months.
Population: Participants who received an allogeneic HSCT while in remission induced by blinatumomab treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 32
percentage of participants | 11.3 [0.0 to 23.4]

12. Secondary Outcome: Serum Blinatumomab Concentration at Steady State
Description: The steady state concentration of blinatumomab was summarized as the observed concentrations collected at least 10 hours after the start of the IV infusion or dose step for cycle 1 and cycle 2, respectively. Serum concentrations of blinatumomab were measured using a validated bioassay. The lower limit of quantitation (LLOQ) = 50.0 pg/mL.
Time Frame: Samples were taken before treatment start and on Days 3, 8, 10, 15, 22, and 29 after infusion start during Cycles 1 and 2.
Population: Pharmacokinetic Data Set (PKS) defined as all patients who received any infusion of blinatumomab and had at least one PK sample collected unless significant protocol deviations affected the data analysis or if key dosing, dosing interruption or sampling information was missing.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Cycle 1: Blinatumomab 9 μg/Day: Participants receiving 9 μg/day blinatumomab by continuous intravenous (CIV) infusion during Cycle 1.
- Cycle 1: Blinatumomab 28 μg/Day: Participants receiving 28 μg/day blinatumomab by continuous intravenous (CIV) infusion during Cycle 1.
- Cycle 2: Blinatumomab 28 μg/Day: Participants receiving 28 μg/day blinatumomab by continuous intravenous (CIV) infusion during Cycle 2.
Arm/Group | Cycle 1: Blinatumomab 9 μg/Day | Cycle 1: Blinatumomab 28 μg/Day | Cycle 2: Blinatumomab 28 μg/Day
Number analyzed (Participants) | 132 | 160 | 88
pg/mL | 211 (258) | 621 (502) | 731 (444)

13. Secondary Outcome: Serum Cytokine Peak Levels
Description: The activation of immune effector cells was monitored by the measurement of peripheral blood cytokine levels including interleukin (IL)-2, IL-4, IL-6, IL-10, tumor necrosis factor (TNF)-α and interferon gamma (IFN)-γ using enzyme-linked immunosorbent assays or cytometric bead assays. The limit of detection of the assay (LOD) was 20 pg/mL and the limit of quantification (LOQ) was 125 pg/mL. Data below LOD were set to 10 pg/mL while data < LOQ and > LOD were reported as measured.
  Serum IL-4 levels were below detection limit (< 20 pg/mL) at all time points in all participants studied.
Time Frame: Serum samples were collected on Days 1 and 8 at 2 hours and 6 hours after treatment start, and on Day 2 (24 hours) and Day 3 (48 hours) of each treatment cycle and on Days 9 and 10 after dose step.
Population: Pharmacodynamic Data Set (PDS): All patients who received any infusion of blinatumomab and had at least one pharmacodynamic sample collected. N indicates the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 189
pg/mL
  IFN-Ɣ: Cycle 1 Week 1 (N=184) | 93.1 (409)
  IFN-Ɣ: Cycle 1 Week 2 (N=175) | 27.4 (83.1)
  IFN-Ɣ: Cycle 2 Week 1 (N=95) | 22.8 (45.8)
  IFN-Ɣ: Cycle 3 Week 1 (N=41) | 21.6 (27.6)
  IL-10: Cycle 1 Week 1 (N=184) | 589 (822)
  IL-10: Cycle 1 Week 2 (N=175) | 95.7 (136)
  IL-10: Cycle 2 Week 1 (N=95) | 397 (633)
  IL-10: Cycle 3 Week 1 (N=41) | 428 (941)
  IL-2: Cycle 1 Week 1 (N=184) | 24.7 (44.6)
  IL-2: Cycle 1 Week 2 (N=175) | 10.8 (5.21)
  IL-2: Cycle 2 Week 1 (N=95) | 11 (5.17)
  IL-2: Cycle 3 Week 1 (N=41) | 10.3 (2.03)
  IL-6: Cycle 1 Week 1 (N=184) | 826 (2390)
  IL-6: Cycle 1 Week 2 (N=175) | 234 (681)
  IL-6: Cycle 2 Week 1 (N=95) | 315 (952)
  IL-6: Cycle 3 Week 1 (N=41) | 69.2 (114)
  TNF-α: Cycle 1 Week 1 (N=184) | 30 (125)
  TNF-α: Cycle 1 Week 2 (N=175) | 10.3 (3.33)
  TNF-α: Cycle 2 Week 1 (N=95) | 12.1 (15)
  TNF-α: Cycle 3 Week 1 (N=41) | 12 (7.79)

14. Secondary Outcome: Percentage of Participants With a Best Response of Blast Free Hypoplastic or Aplastic Bone Marrow Within 2 Cycles of Treatment
Description: Blast Free Hypoplastic or Aplastic Bone Marrow was defined as:
  * bone marrow blasts ≤ 5%
  * no evidence of disease
  * insufficient recovery of peripheral counts: platelets ≤ 50,000/μL and/or absolute neutrophil count (ANC) ≤ 500/μL
Time Frame: Within the first 2 cycles of treatment, 12 weeks
Population: Primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 189
percentage of participants | 9.0 [5.3 to 14.0]

15. Secondary Outcome: Best Response During the Core Study
Description: Complete Remission (CR):
  * bone marrow blasts ≤ 5%
  * no evidence of disease
  * full recovery of peripheral blood counts:
    * platelets > 100,000/μL, and
    * absolute neutrophil count (ANC) > 1,000/μL
  Complete Remission With Partial Hematological Recovery (CRh*):
  * bone marrow blasts ≤ 5%
  * no evidence of disease
  * partial recovery of peripheral blood counts:
    * platelets > 50,000/μL, and
    * ANC > 500/μL
  Blast Free Hypoplastic or Aplastic Bone Marrow:
  * bone marrow blasts ≤ 5%
  * no evidence of disease
  * insufficient recovery of peripheral counts: platelets ≤ 50,000/μL and/or ANC ≤ 500/μL
  Partial Remission:
  • bone marrow blasts 6% to 25% with at least a 50% reduction from Baseline.
Time Frame: From the first dose of blinatumomab until 30 days after the end of the last infusion during the core study, or until the data cut-off date of 10 October 2013; a maximum of 7.5 months.
Population: Primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 189
percentage of participants
  Remission (CR/CRh*) | 43.4 [36.2 to 50.8]
  Complete Remission | 35.4 [28.6 to 42.7]
  Complete remission with only partial hematological | 7.9 [4.5 to 12.8]
  Blast free hypoplastic or aplastic bone marrow | 9.0 [5.3 to 14.0]
  Partial remission | 2.6 [0.9 to 6.1]

ADVERSE EVENTS:
Time Frame: From the start of the first infusion to 30 days after the end of the last infusion in the core study or from the start of the first retreatment cycle infusion to 30 days after the end of the last retreatment cycle, median treatment duration was 42.2 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Blinatumomab: Participants received blinatumomab by continuous intravenous (CIV) infusion over 4 weeks followed by a treatment-free interval of 2 weeks for up to 5 consecutive cycles. The the initial dose was 9 μg/day for the first seven days of treatment, escalated to 28 μg/day starting from Week 2 of treatment.
Arm/Group | Blinatumomab
Serious Adverse Events (participants affected / at risk) | 121/189
Other Adverse Events (participants affected / at risk) | 186/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=189)
Anaemia (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 16
Leukocytosis (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 7
Pancytopenia (Blood and lymphatic system disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Aplasia (Congenital, familial and genetic disorders) | 1
Diplopia (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Chest pain (General disorders) | 2
Device occlusion (General disorders) | 2
Disease progression (General disorders) | 3
Fatigue (General disorders) | 1
Hypothermia (General disorders) | 1
Medical device complication (General disorders) | 3
Mucosal inflammation (General disorders) | 1
Multi-organ failure (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 11
Cytokine release syndrome (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Abdominal infection (Infections and infestations) | 1
Aspergillus infection (Infections and infestations) | 2
BK virus infection (Infections and infestations) | 1
Bacterial sepsis (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Candida infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Cholecystitis infective (Infections and infestations) | 1
Device related infection (Infections and infestations) | 7
Enterobacter infection (Infections and infestations) | 1
Enterococcal bacteraemia (Infections and infestations) | 2
Enterococcal infection (Infections and infestations) | 2
Enterococcal sepsis (Infections and infestations) | 2
Epididymal infection (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 2
Fungal infection (Infections and infestations) | 2
Fusarium infection (Infections and infestations) | 2
Gastrointestinal infection (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 4
Kidney infection (Infections and infestations) | 1
Klebsiella infection (Infections and infestations) | 1
Leuconostoc infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 2
Pathogen resistance (Infections and infestations) | 1
Pilonidal cyst (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 9
Pneumonia fungal (Infections and infestations) | 2
Pneumonia klebsiella (Infections and infestations) | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1
Pseudomonal bacteraemia (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Pulmonary sepsis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 9
Septic shock (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 1
Sinusitis fungal (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 4
Staphylococcal infection (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 2
Streptococcal sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Viral haemorrhagic cystitis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 5
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 3
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
C-reactive protein increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Fistula (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 2
Ataxia (Nervous system disorders) | 3
Cerebral haemorrhage (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 3
Convulsion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 5
Headache (Nervous system disorders) | 4
Hemiparesis (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 1
Neurotoxicity (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 1
Poor quality sleep (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 5
Trigeminal nerve disorder (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 5
Delirium febrile (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Bladder perforation (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Scrotal oedema (Reproductive system and breast disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Catheter placement (Surgical and medical procedures) | 2
Central venous catheter removal (Surgical and medical procedures) | 1
Resuscitation (Surgical and medical procedures) | 1
Capillary leak syndrome (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Femoral artery occlusion (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Hypovolaemic shock (Vascular disorders) | 1
Subclavian vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=189)
Anaemia (Blood and lymphatic system disorders) | 37
Febrile neutropenia (Blood and lymphatic system disorders) | 38
Leukopenia (Blood and lymphatic system disorders) | 19
Neutropenia (Blood and lymphatic system disorders) | 26
Thrombocytopenia (Blood and lymphatic system disorders) | 21
Sinus tachycardia (Cardiac disorders) | 11
Tachycardia (Cardiac disorders) | 11
Vision blurred (Eye disorders) | 12
Abdominal distension (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 31
Abdominal pain upper (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 39
Diarrhoea (Gastrointestinal disorders) | 34
Nausea (Gastrointestinal disorders) | 46
Vomiting (Gastrointestinal disorders) | 25
Asthenia (General disorders) | 17
Chest pain (General disorders) | 19
Chills (General disorders) | 29
Fatigue (General disorders) | 28
Oedema (General disorders) | 11
Oedema peripheral (General disorders) | 49
Pain (General disorders) | 14
Pyrexia (General disorders) | 106
Cytokine release syndrome (Immune system disorders) | 22
Upper respiratory tract infection (Infections and infestations) | 10
Alanine aminotransferase increased (Investigations) | 23
Aspartate aminotransferase increased (Investigations) | 20
Blood bilirubin increased (Investigations) | 12
Immunoglobulins decreased (Investigations) | 17
Weight increased (Investigations) | 16
Decreased appetite (Metabolism and nutrition disorders) | 19
Hyperglycaemia (Metabolism and nutrition disorders) | 23
Hypokalaemia (Metabolism and nutrition disorders) | 44
Hypomagnesaemia (Metabolism and nutrition disorders) | 25
Hypophosphataemia (Metabolism and nutrition disorders) | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 18
Back pain (Musculoskeletal and connective tissue disorders) | 25
Bone pain (Musculoskeletal and connective tissue disorders) | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10
Muscular weakness (Musculoskeletal and connective tissue disorders) | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20
Dizziness (Nervous system disorders) | 25
Headache (Nervous system disorders) | 63
Tremor (Nervous system disorders) | 33
Anxiety (Psychiatric disorders) | 14
Insomnia (Psychiatric disorders) | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 35
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11
Petechiae (Skin and subcutaneous tissue disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 22
Hypertension (Vascular disorders) | 12
Hypotension (Vascular disorders) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.